CLINICAL TRIAL: NCT05350514
Title: Preclinical Imaging Biomarkers of Alzheimer's Disease Neuropathology in Young Adults With Youth-onset Diabetes: a Proof-of-concept Study
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American College of Radiology (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0608
Record Dates: First submitted 2022-04-12; First posted 2022-04-28 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Youth Onset
Keywords: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Youth Onset; Magnetic Resonance Imaging; Positron Emission Tomography Imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T1D: Young adults with youth-onset type 1 diabetes (n=5) from the SEARCH for Diabetes in Youth study cohort
  Interventions: Drug: PI-2620 tracer
- T2D: Young adults with youth-onset type 2 diabetes (n=5) from the SEARCH for Diabetes in Youth study cohort
  Interventions: Drug: PI-2620 tracer
- NDM: Age-similar group of young adults without diabetes (n=5)
  Interventions: Drug: PI-2620 tracer

INTERVENTIONS:
Drug: PI-2620 tracer — Following published manufacturer guidelines for Flutemetamol (VizamylTM), Flortaucipir (TauvidTM) and PI-2620 tracer administration162, all participants will be given a 370 MBq (10 mCi) single intravenous bolus (total volume 10mL) of the radiotracer, followed with an intravenous flush of 0.9% sodium chloride injection. Radiotracer administration and participant monitoring will be conducted by trained personnel from the CU-RIC.

SUMMARY:
The goal of the study is to characterize preclinical Alzheimer's Disease and related dementias (AD/ADRD) neuropathology in a selected group of young adults with youth-onset diabetes, and an age-similar group of young adults without diabetes.

DETAILED DESCRIPTION:
The goal of the current proof-of-concept study is to characterize brain structural, functional, and molecular imaging biomarkers of preclinical Alzheimer's Disease and related dementias (AD/ADRD) neuropathology in a selected group of young adults with youth-onset diabetes (Y-DM; type 1 diabetes [T1D], n=5; type 2 diabetes [T2D], n=5) from the SEARCH for Diabetes in Youth study cohort, and an age-similar group of young adults without diabetes (n=5). This study will quantify structural and functional imaging biomarkers of AD/ADRD neuropathology via magnetic resonance imaging by assessing gray matter (GM) volume/cortical thickness, as well as GM and white matter (WM) microstructure, resting state functional network connectivity (rsfMRI), and cerebral blood flow (CBF) and WM hyperintensity volume. This study will additionally quantify brain tau density via positron emission tomography as the gold-standard measure of preclinical AD/ADRD neuropathology.

ELIGIBILITY:
Inclusion Criteria:

* Part of the SEARCH for Diabetes in Youth study cohort or
* Age 18-40
* Without diabetes

Exclusion Criteria:

* Head trauma with loss of consciousness >30 minutes
* Claustrophobia
* Metal in the body
* Major psychiatric disorder (eg. schizophrenia, bipolar, and major depression)
* Neurological conditions affecting cognition (eg. epilepsy)
* Stroke
* If female, breastfeeding, plan to become pregnant or are pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of young adults with youth-onset type 1 diabetes and type 2 diabetes from the SEARCH for Diabetes in Youth study cohort, and an age-similar group of young adults (18-40 years old) without diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Temporal lobe volume in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Voxel-based morphometry via Sagittal 3D Accelerated MPRAGE/IRSPGR
Temporal lobe cortical thickness in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Voxel-based morphometry via Sagittal 3D Accelerated MPRAGE/IRSPGR
Whole brain white matter hyperintensities volume in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Structural cerebrovascular disease via Sagittal 3D FLAIR
Regional homogeneity of the default mode network in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Resting-state functional connectivity via Axial T2* EPI fcMRI
Whole brain cerebral blood flow in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Cerebral blood flow or perfusion via Axial 3D pCASL
Whole brain fractional anisotropy in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Gray matter and white matter microstructure via Diffusion Kurtosis Imaging
Standardized uptake value ratio for hippocampal to cerebellar comparison in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Tau accumulation via positron emission tomography with PI-2620 radiotracer
Standardized uptake value ratio for entorhinal to cerebellar comparison in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Tau accumulation via positron emission tomography with PI-2620 radiotracer
Standardized uptake value ratio for cerebral to cerebellar comparison in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Tau accumulation via positron emission tomography with PI-2620 radiotracer

SECONDARY OUTCOMES:
Whole brain gray matter volume in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Voxel-based morphometry via Sagittal 3D Accelerated MPRAGE/IRSPGR
Whole brain white matter volume in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Voxel-based morphometry via Sagittal 3D Accelerated MPRAGE/IRSPGR
Perivascular space in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Structural cerebrovascular disease via Sagittal 3D FLAIR
Atlas based region of interest cerebral blood flow in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Cerebral blood flow via Axial 3D pCASL
Atlas based region of interest fractional anisotropy in young adults with Type 1 diabetes, Type 2 diabetes, and young adults without diabetes | Baseline
  Gray matter and white matter microstructure via Diffusion Kurtosis Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Allison Shapiro, PhD, MPH, Principal Investigator — University of Colorado, Denver; Christopher T Whitlow, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Lifecourse Epidemiology of Adiposity and Diabetes Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No